CLINICAL TRIAL: NCT00309881
Title: CHOP Plus Rituximab (CHOP-R) in Fludarabine Refractory Chronic Lymphocytic Leukemia (CLL) or CLL With Autoimmune Haemolytic Anemia (AIHA) or Richter's Transformation (RT)
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Chronic Lymphocytic Leukemia (CLL) That Did Not Respond to Fludarabine, CLL With Autoimmune Haemolytic Anemia (AIHA) or Richter's Transformation (RT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CLL2G; EU-20549; GCLLSG-423; MEDAC-GCLLSG-CLL2G
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving more than one drug (combination chemotherapy) together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with rituximab works in treating patients with chronic lymphocytic leukemia (CLL) that has not responded to fludarabine (closed to entry as of 10/2006), CLL with autoimmune hemolytic anemia, or Richter transformation.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy, in terms of the rate and quality of remission, of chemotherapy comprising cyclophosphamide, doxorubicin hydrochloride, vincristine, prednisone, and rituximab (CHOP-R) in patients with fludarabine-refractory chronic lymphocytic leukemia (CLL) (closed to accrual as of 10/2006), CLL with autoimmune hemolytic anemia, or Richter transformation.
* Determine the incidence of infection in patients on CHOP-R regimen.

Secondary

* Determine the toxicity of this regimen in these patients
* Determine the progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is a prospective, multicenter study. Patients are stratified according to disease (chronic lymphocytic leukemia (CLL) (closed to accrual as of 10/2006) vs CLL with autoimmune hemolytic anemia vs Richter transformation).

Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Patients also receive rituximab IV on day 1 of the second course and each subsequent course. Treatment repeats every 21 days for up to 6 (for patients with CLL) or 8 (for patients with Richter's transformation) courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of previously treated chronic lymphocytic leukemia (CLL) meeting the following criteria:

  * Binet stage B (Rai stages I and II) or Binet stage C (Rai stages III and IV) disease
  * Rapid disease progression, symptomatic enlarged lymph nodes, or severe B-cell symptoms
* CLL with autoimmune hemolytic anemia allowed
* Richter transformation allowed

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months
* ECOG performance status 0-3
* No severe organ dysfunction
* No other prior or concurrent neoplasms

PRIOR CONCURRENT THERAPY:

* No more than 4 prior chemotherapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2003-04; Primary Completion 2006-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Rate of remission
Quality of remission

SECONDARY OUTCOMES:
Toxicity
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (18):
- Germany (18):
  - Kreiskrankenhaus, Bad Hersfeld
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Universitaetsklinikum Essen, Essen
  - Gemeinschaftspraxis Fuer Innere Medizin, Hematologie Und Onkologie, Giessen
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Allgemeines Krankenhaus Hagen, Hagen
  - Praxis fur Innere Medizin - Hamburg, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Marienhospital at Ruhr University Bochum, Herne
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Oldenburg, Oldenburg
  - Marienhospital Stuttgart, Stuttgart
  - Haematologische Praxis, Weiden
  - Medizinische Poliklinik, Universitaet Wuerzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Langerbeins P, Busch R, Anheier N, Durig J, Bergmann M, Goebeler ME, Hurtz HJ, Stauch MB, Stilgenbauer S, Dohner H, Fink AM, Cramer P, Fischer K, Wendtner CM, Hallek M, Eichhorst B. Poor efficacy and tolerability of R-CHOP in relapsed/refractory chronic lymphocytic leukemia and Richter transformation. Am J Hematol. 2014 Dec;89(12):E239-43. doi: 10.1002/ajh.23841. Epub 2014 Sep 26. PMID 25196783